CLINICAL TRIAL: NCT03542994
Title: A Phase 1a/1b Randomized Double-blind Placebo-controlled Single and Multiple Ascending Dose Study of EDP1066 in Healthy Participants and Participants With Mild to Moderate Psoriasis and Atopic Dermatitis
Brief Title: A Study of EDP1066 in Healthy Participants and Participants With Mild to Moderate Psoriasis and Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: EDP1066-001; 2017-004337-90 (EudraCT Number)
Record Dates: First submitted 2018-04-24; First posted 2018-06-01 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Psoriasis; Atopic Dermatitis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: The study is a double-blind dose escalation cohort study in healthy volunteers and participants with either mild to moderate psoriasis or mild to moderate atopic dermatitis. The study consists of 9 cohorts and will test doses of EDP1066 versus placebo. The safety and tolerability of EDP1066 will be tested in participants with psoriasis and atopic dermatitis alongside pharmacodynamic effects on the systemic immune system and observation of any clinical effects.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Other): 12 healthy volunteers; 8 on EDP1066, 4 on placebo. Dose=up to a maximum of 66 mg, capsule, once daily, 15 days
  Interventions: Other: EDP1066; Drug: Placebo oral capsule
- Cohort 2 (Other): 12 healthy volunteers; 8 on EDP1066, 4 on placebo. Dose=up to a maximum of 660 mg, capsule, once daily, 15 days
  Interventions: Other: EDP1066; Drug: Placebo oral capsule
- Cohort 3 (Other): 12 healthy volunteers; 8 on EDP1066, 4 on placebo. Dose=up to a maximum of 3.3 g, capsule, once daily, 15 days
  Interventions: Other: EDP1066; Drug: Placebo oral capsule
- Cohort 4 (Other): 12 subjects with mild to moderate psoriasis; 8 on EDP1066, 4 on placebo. Dose=up to a maximum of 660 mg, capsule, once daily, 29 days
  Interventions: Other: EDP1066; Drug: Placebo oral capsule
- Cohort 5 (Other): 24 subjects with mild to moderate psoriasis; 16 on EDP1066, 8 on placebo. Dose=up to a maximum of 3.3 g, capsule, once daily, 29 days
  Interventions: Other: EDP1066; Drug: Placebo oral capsule
- Cohort 6 (Other): up to 24 subjects with mild to moderate atopic dermatitis; 16 on EDP1066, 8 on placebo.
  Dose=up to a maximum of 660 mg, capsule, once daily, 29 days
  Interventions: Other: EDP1066; Drug: Placebo oral capsule
- Cohort 7 (Other): up to 24 subjects with mild to moderate atopic dermatitis; 16 on EDP1066, 8 on placebo.
  Dose=up to a maximum of 3.3 g, capsule, once daily, 29 days
  Interventions: Other: EDP1066; Drug: Placebo oral capsule
- Cohort 8 (Other): up to 24 subjects with mild to moderate psoriasis; 16 on EDP1066, 8 on placebo. Dose=up to a maximum of 3.3g, capsule, once daily, 29 days
  Interventions: Other: EDP1066; Drug: Placebo oral capsule
- Cohort 9 (Other): up to 24 subjects with mild to moderate atopic dermatitis; 16 on EDP1066, 8 on placebo.
  Dose=up to a maximum of 3.3 g, capsule, once daily, 29 days
  Interventions: Other: EDP1066; Drug: Placebo oral capsule

INTERVENTIONS:
Other: EDP1066 — EDP1066 is an orally administered monoclonal microbial
Drug: Placebo oral capsule — placebo

SUMMARY:
Evelo will investigate the safety and tolerability of EDP1066 and its potential to be a medicinal product in healthy volunteers and individuals with mild to moderate psoriasis and atopic dermatitis.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled clinical study with dose escalations to assess safety, tolerability, and pharmacodynamic effect of EDP1066. Since this clinical study is the first study in humans, the participants will be healthy volunteers or subjects with mild to moderate psoriasis or atopic dermatitis who are otherwise well. Investigation of EDP1066 in this patient population provides an opportunity to gain pharmacodynamic information using a range of tissue biopsies and composite clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

General:

* Participant has a body mass index of ≥ 18 kg/m2 to ≤ 35 kg/m2 at Screening.

Healthy Volunteers:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.

Mild to moderate psoriasis:

1. Participant has had a confirmed diagnosis of mild to moderate plaque-type psoriasis for at least 6 months involving ≤ 5% of body surface area (BSA) (excluding the scalp).
2. Participant has a minimum of 2 psoriatic lesions with at least 1 plaque in a site suitable for biopsy.

Mild to moderate atopic dermatitis:

1. Mild to moderate atopic dermatitis with a minimum of 3% to a maximum of 15% BSA involvement.
2. Participant has had a confirmed diagnosis of mild to moderate atopic dermatitis for at least 6 months IGA score of 2 or 3.
3. Participant has a minimum of 2 atopic dermatitis lesions with at least 1 in a site suitable for biopsy.

Exclusion Criteria:

1. Female participant who is pregnant, or plans to become pregnant during the study, or breastfeeding, or sexually active with childbearing potential who is not using a medically accepted birth control method.
2. Participant has received live attenuated vaccination within 6 weeks prior to Screening or intends to have such a vaccination during the course of the study.
3. Participant has received any investigational drug or experimental procedure within 90 days or 5 half-lives, whichever is longer, prior to study intervention administration.
4. Participant requires treatment with an anti-inflammatory drug during the study period. Paracetamol will be permitted for use as an antipyretic and/or analgesic (maximum of 2 grams/day in any 24 hour period).
5. Participant has an active infection (e.g. sepsis, pneumonia, abscess) or has had an infection requiring antibiotic treatment within 6 weeks prior to Investigational Medicinal Product (IMP) administration. When in doubt, the investigator should confer with the Sponsor study physician.
6. Participant has renal or liver impairment, defined as:

   a. For healthy volunteers: i. For women, serum creatinine level ≥ 125 μmol/L; for men, ≥ 135 μmol/L, or ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 1.5 x upper limit of normal (ULN), or iii. Alkaline phosphatase (ALP) and/or bilirubin > 1.5 x ULN b. For participants with mild to moderate atopic dermatitis or psoriasis: i. For women, serum creatinine level ≥ 125 μmol/L; for men, ≥ 135 μmol/L, or ii. ALT or AST > 2 x ULN and/or bilirubin > 1.5 x ULN

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measured through Adverse Events (AEs) | Day 1 to Day 60
  Number of participants with AEs by seriousness and relationship to treatment
Safety and tolerability measured through lab measurements | Day 0 to Day 60
  Number of participants with clinically significant change from baseline (Day 0) in laboratory values
Safety and tolerability measured through ECG | Day 0 to Day 60
  Number of participants with clinically relevant changes from baseline (Day 0) ECG parameters
Safety and tolerability measured through physical examination | Day 1 to Day 60
  Physical examination of stool samples based on the Bristol Stool Scale (Types 3 and 4 are ideal stool):
  Type 1: Separate hard lumps, like nuts (hard to pass); Type 2: Sausage-shaped, but lumpy; Type 3: Like a sausage but with cracks on its surface; Type 4: Like a sausage or snake, smooth and soft; Type 5: Soft blobs with clear cut edges (easy to pass); Type 6: Fluffy pieces with ragged edges, a mushy stool; Type 7: Watery, no solid pieces, entirely liquid
GI safety measurement through biomarker analysis | Day 1 to Day 60
  GI safety measurement through fecal calprotectin analysis

SECONDARY OUTCOMES:
Clinical improvement in subjects with mild to moderate psoriasis | Day 0 to Day 60
  Change from baseline (Day 0) Psoriasis-area-and-severity index score (PASI) in response to EDP1066, measured on a scale of 0 to 6 (where 0 is most favorable and 6 is least favorable).
Clinical improvement in subjects with mild to moderate atopic dermatitis | Day 0 to Day 60
  Change from baseline (Day 0) Eczema-area-and-severity index score (EASI) in response to EDP1066, measured on a scale of 0 to 6 (where 0 is most favorable and 6 is least favorable).

CONTACTS AND LOCATIONS:
Overall Officials: Duncan McHale, MD, PhD, Study Director — Evelo Biosciences; Daryl Bendel, MBChB, MBA, Principal Investigator — University of Surrey; Giuseppe Fiore, MD, Principal Investigator — Medicines Evaluation Unit Ltd; Aliya Asher, MD, Principal Investigator — MAC Clinical Research; Richard Fitzgerald, MD, Principal Investigator — Royal Liverpool Hospital
Locations (7):
- United Kingdom (7):
  - University of Surrey Clinical Research Center, Guildford, Surrey
  - MAC Clinical Research, Barnsley
  - MAC Clinical Research, Cannock
  - Royal Liverpool Clinical Research Unit, Liverpool
  - MAC Clinical Research, Manchester
  - Medicines Evaluation Unit Ltd., The Langley Building, Wythenshawe Hospital, Manchester
  - MAC Clinical Research, Stockton-on-Tees